CLINICAL TRIAL: NCT07126483
Title: A Randomized Controlled Non-Inferiority Trial Comparing Thoracic Paravertebral Block and Intrathecal Morphine for Postoperative Analgesia in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: Thoracic Paravertebral Block vs Intrathecal Morphine in VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, Prof. Dr., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITMTPVB2025
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Acute Pain; Video-Assisted Thoracoscopic Surgery; Intrathechal Morphine; Paravertebral Peripheral Nerve Block
Keywords: Thoracic Paravertebral Block; Intrathecal Morphine;; Video-Assisted Thoracoscopic Surgery; Postoperative Analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Paravertebral Block (TPVB) (Experimental): Patients in this group will receive a single-injection ultrasound-guided thoracic paravertebral block before induction of standardized general anesthesia. The block will be performed using 0.4 mL/kg of 0.25% bupivacaine with epinephrine (1:400,000). Postoperatively, patients will receive intravenous patient-controlled analgesia with morphine, along with scheduled paracetamol and NSAIDs.
  Interventions: Procedure: Thoracic paravertebral block
- Intrathecal Morphine (ITM) (Experimental): Patients in this group will receive a single dose of intrathecal morphine (5 mcg/kg diluted in 3 mL 0.9% saline) at the L3-L4 or L4-L5 interspace before induction of standardized general anesthesia. Postoperatively, patients will receive intravenous patient-controlled analgesia with morphine, along with scheduled paracetamol and NSAIDs.
  Interventions: Drug: Morphine

INTERVENTIONS:
Procedure: Thoracic paravertebral block — Ultrasound-guided single-injection thoracic paravertebral block using 0.4 mL/kg of 0.25% bupivacaine with epinephrine (1:400,000) before induction of standardized general anesthesia. Postoperative analgesia will be provided with intravenous patient-controlled analgesia morphine, along with scheduled paracetamol and NSAIDs.
  Other Names: TPVB
  Arms: Thoracic Paravertebral Block (TPVB)
Drug: Morphine — Single intrathecal injection of morphine (5 mcg/kg diluted in 3 mL 0.9% saline) at the L3-L4 or L4-L5 interspace before induction of standardized general anesthesia. Postoperative analgesia will be provided with intravenous patient-controlled analgesia morphine, along with scheduled paracetamol and NSAIDs.
  Other Names: Intrathecal Morphine (ITM)
  Arms: Intrathecal Morphine (ITM)

SUMMARY:
The purpose of this study is to find out which pain relief method works better for people having video-assisted thoracoscopic surgery. We will compare two techniques: thoracic paravertebral block (TPVB), a numbing injection near the spine, and intrathecal morphine (ITM), a small dose of morphine injected into the spinal fluid. We want to see if ITM works as well as TPVB in reducing the need for pain medicine during the first 24 hours after surgery. People in the study will get either TPVB or ITM before going to sleep for surgery, use a patient-controlled pain pump after surgery, and have their pain scores, medicine use, recovery, and possible side effects checked for up to 30 days after surgery.

DETAILED DESCRIPTION:
This study will compare two different pain control techniques for people having video-assisted thoracoscopic surgery (VATS), a minimally invasive chest operation. The first technique, called thoracic paravertebral block (TPVB), involves injecting numbing medicine near the spine to block pain from the surgical area. The second technique, intrathecal morphine (ITM), involves giving a small dose of morphine into the spinal fluid to provide pain relief after surgery.

The main goal is to find out if ITM works as well as TPVB in reducing the need for additional pain medicine during the first 24 hours after surgery. This is a randomized controlled trial, meaning participants will be randomly assigned to one of the two groups. Everyone will receive general anesthesia for their surgery and will use a patient-controlled analgesia pump afterwards, along with regular pain medicines such as paracetamol and tenoxicam.

Pain scores, the amount of pain medicine used, and recovery quality will be measured at regular times in the first 24 hours after surgery. We will also monitor side effects such as nausea, vomiting, itching, or breathing problems. All patients will be followed for 30 days after surgery to check for any complications.

ELIGIBILITY:
Inclusion Criteria

1. Age between 18 and 75 years
2. American Society of Anesthesiologists (ASA) physical status I-III
3. Scheduled for elective video-assisted thoracoscopic surgery (VATS) for wedge resection, segmentectomy, or lobectomy
4. Ability to understand the study protocol and provide written informed consent

Exclusion Criteria

1. Refusal to participate
2. Pregnancy
3. Morbid obesity (body mass index > 30)
4. Known allergy to opioids, local anesthetics, or NSAIDs
5. History of neuropsychiatric disorder, cognitive impairment, or inability to communicate with investigators
6. History of substance abuse
7. Current anticoagulant use or known bleeding disorder
8. Presence of systemic infection
9. Significant cardiovascular, hepatic, renal, or endocrine disease
10. History of chronic pain syndromes or chronic pain treatment
11. Emergency surgery or previous ipsilateral VATS or thoracotomy
12. Preoperative chronic opioid therapy within 3 months (≥15 mg/day for ≥30 days)
13. Severe intraoperative or postoperative bleeding, hemodynamic instability
14. Requirement for prolonged postoperative ventilation (> 18 hours)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Cumulative IV Morphine Milligram Equivalents (IV-MME) in the First 24 Hours After Surgery | First 24 hours postoperatively
  Total amount of intravenous morphine milligram equivalents (IV-MME) administered during the first 24 postoperative hours.

SECONDARY OUTCOMES:
Cumulative IV Morphine Milligram Equivalents (IV-MME) in the First 12 Hours After Surgery | First 12 hours postoperatively
  Total amount of IV-MME administered during the first 12 postoperative hours.
Time to First Analgesic Request | From extubation and recovery of communication ability to first PCA demand, within 24 hours postoperatively
  Duration from the time the patient is extubated and able to communicate after surgery to the first patient-controlled analgesia (PCA) demand for analgesia
Numeric Rating Scale (NRS) Pain Scores at Rest | 0, 3, 6, 12, 18, and 24 hours postoperatively
  Pain intensity at rest measured using an 11-point NRS (0 = no pain, 10 = worst pain imaginable) at 0, 3, 6, 12, 18, and 24 hours postoperatively.
Numeric Rating Scale (NRS) Pain Scores During Coughing or Deep Breathing | 0, 3, 6, 12, 18, and 24 hours postoperatively
  Pain intensity during coughing or deep breathing measured using an 11-point NRS (0 = no pain, 10 = worst pain imaginable) at 0, 3, 6, 12, 18, and 24 hours postoperatively.
Sedation Score | 0, 3, 6, 12, 18, and 24 hours postoperatively
  Sedation Score assessed using the Ramsay Sedation Scale (1-6) at 0, 3, 6, 12, 18, and 24 hours postoperatively
Postoperative Nausea and Vomiting (PONV) Score | 0, 3, 6, 12, 18, and 24 hours postoperatively
  Score of PONV, assessed using a 4-point scale (0 = none, 1 = nausea only, 2 = single episode of vomiting, 3 = multiple episodes of vomiting).
Pruritus Score | 0, 3, 6, 12, 18, and 24 hours postoperatively
  Score of pruritus, assessed using a 4-point scale (0-3; 0 none, 1 mild/no treatment, 2 moderate/treatment, 3 severe/repeat treatment; treatment threshold ≥2)
Rescue Analgesia Requirement | First 24 hours postoperatively
  Number of participants requiring additional analgesics beyond PCA during the first 24 hours postoperatively.
Incidence of Postoperative Complications | First 30 postoperative days
  Number of participants experiencing any postoperative complication within 30 days
Quality of Recovery questionnaire (QoR-15) score | Preoperative baseline (≤24 h before surgery), 24 h postoperatively, and at hospital discharge (anticipated within 3 days)
  Recovery quality wil be assessed with the validated Turkish QoR-15 (15 items; total 0-150, higher scores = better recovery).
Intraoperative Remifentanil and Propofol Consumption | Intraoperative period (from induction to 240 min)
  Total intraoperative doses of remifentanil and propofol administered by the anesthesia team will be recorded.
Intraoperative Hemodynamics (Heart Rate and Mean Arterial Pressure) | Intraoperative period (from induction to 240 min)
  Heart rate and mean arterial pressure will be recorded at standard clinical intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including baseline characteristics, intraoperative and postoperative outcome measures, and adverse events) will be shared with researchers upon reasonable request for academic purposes. Data will be available beginning 6 months after publication of the primary results and for up to 5 years. Access will be granted following approval of a written proposal and data use agreement.
Supporting Information: Study Protocol, SAP, ICF